CLINICAL TRIAL: NCT05160155
Title: Comparison of the Analgesic Efficacy of Serratus Anterior Plane Block and Intercostal Block for Rib Fractures
Brief Title: Comparison of the Analgesic Efficacy of Serratus Anterior Plane Block and Intercostal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-21-2143
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Rib Fractures; Serratus Anterior Plane Block; Erector Spinae Plane Block; Acute Pain
Keywords: Rib Fractures; Serratus Anterior Plane Block; Erector Spinae Plane Block
MeSH Terms: conditions — Rib Fractures; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Anterior Plane Block (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique above the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine will be injected into the area. The block will be terminated.
  Interventions: Procedure: Serratus Anterior Plane Block
- Intercostal Block (Active Comparator): The USG probe will be placed at the level of the posterior axillary line and the broken ribs. The ribs, external intercostal muscle, and internal intercostal muscle structures will be imaged. 3 ml of 0.25% bupivacaine will be injected into the subcostal area. This 3 ml 0.25% bupivacaine injection will be administered for each broken rib. The block will be terminated.
  Interventions: Procedure: Intercostal Block

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — Serratus anterior plane block will be performed unilaterally, under US guidance.
  Arms: Serratus Anterior Plane Block
Procedure: Intercostal Block — Intercostal Block will be performed unilaterally, under US guidance.
  Arms: Intercostal Block

SUMMARY:
More than 50% of patients presenting with chest trauma experience rib fractures and these rib fractures are associated with significant morbidity, mortality, and long-term disability. Many of these adverse outcomes result from poorly controlled pain that interferes with breathing, leading to atelectasis, pneumonia, and respiratory failure. Therefore, early provision of adequate analgesia is crucial in the management of these patients. The basic stones of analgesic therapy are oral and intravenous drugs such as paracetamol, nonsteroidal anti-inflammatory drugs (NSAIDs), and opioids. However, patients with more significant injuries or comorbidities often require interventional procedures to provide adequate analgesia and avoid opioid-related side effects. Thoracic epidural analgesia and thoracic paravertebral blocks have traditionally been used, but these techniques are associated with side effects and may cause hemodynamic instability. Today, the use of ultrasonography (USG) guided block techniques such as erector spinae plane block (ESPB), serratus anterior plane block (SAPB) and intercostal block (ICB) has increased. These techniques are considered to be simpler and theoretically safer. Although ICB is frequently mentioned in the literature, the publications of new plane blocks such as ESPB and SAPB are new and few in number. In this study, SAPB and ICP to be performed with USG will be evaluated in terms of analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index between 18-30 kg/m2
* Patients with 6 or less rib fractures

Exclusion Criteria:

* Patient refusing the procedure
* History of chronic analgesic or opioid therapy
* History of local anesthetic allergy
* Infection in the intervention area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Pain scores | 24 hours after block
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th and 24th hours after surgery.

SECONDARY OUTCOMES:
Need for additional analgesia | 24 hours after block
  Whether the patients need additional analgesia after the block and the amount of additional analgesia needed will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No